CLINICAL TRIAL: NCT06422377
Title: An Open-label, Nonrandomized, Phase 3 Study to Evaluate the Efficacy and Safety of Soticlestat in Participants With Dravet Syndrome or Lennox-Gastaut Syndrome Who Have Been Exposed to Fenfluramine
Brief Title: A Study Evaluating Soticlestat in Participants With Dravet Syndrome or Lennox-Gastaut Syndrome Who Have Been Exposed to Fenfluramine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision unrelated to patient safety.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-935-3004; 2023-504104-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dravet Syndrome (DS); Lennox-Gastaut Syndrome (LGS)
Keywords: Drug Therapy
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — soticlestat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Soticlestat (Experimental): Participant received soticlestat at a starting dose of 100 mg to 200 mg in the 4-week titration. As a part of maintenance (initially planned for 48 weeks per protocol), participant remained on the 200 mg BID dose for 9 days followed by a 1-week taper to receive soticlestat 100 mg BID.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablets or mini-tablets
  Other Names: TAK-935

SUMMARY:
The purpose of this study is to check how soticlestat impacts symptoms of Dravet syndrome [DS] and Lennox-Gastaut syndrome [LGS] in participants who have been exposed to fenfluramine.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat. Soticlestat is being tested to treat people who have DS or LGS and have been exposed to fenfluramine. This study will assess the efficacy and safety of soticlestat in addition to standard care in the treatment of DS or LGS.

The study will enroll approximately 45 patients. This study comprises a screening period of up to 6 weeks, a 4-week titration period, a 48-week maintenance period, a taper period of up to 1 week and a follow-up safety visit. Participants will be enrolled to receive soticlestat along with the standard of care:

• Soticlestat 100-300 milligrams (mg)

Participants will receive oral administration of soticlestat Dose 1 (days 1 to 7), Dose 2 (days 8 to 14), and Dose 3 (Days 15 to 28) with a minimum dose of 100 mg to a maximum dose of 300 mg depending on participant's body weight in the titration period followed by maintenance period up to end of treatment (up to approximately 52 weeks). Percent change from baseline in convulsive in participants with DS and major motor drop (MMD) in participants with LGS seizure frequency per 28 days during the initial 12 weeks of the maintenance period will be assessed.

This multi-center trial will be conducted in the United Kingdom and Europe. The overall time to participate in this study is approximately 60 weeks. Participants will make multiple visits to the clinic and will be followed up for safety by visiting the clinic or by telephone approximately 2 weeks after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has been exposed to fenfluramine (currently on or used previously).
2. The participant has a clinical diagnosis of LGS and a history of, on average, ≥12 MMD seizures in the last 90 days immediately before screening based on historical information, and the participant has ≥4 MMD seizures during a minimum of 4 weeks of seizure data collection during the prospective baseline period.
3. The participant is currently taking 0 to 5 antiseizure treatments (eg. antiseizure medications [ASMs], vagus nerve stimulation [VNS], ketogenic diet) at stable doses.

Exclusion Criteria:

1. The participant is currently enrolled in a clinical study involving an investigational product or treatment device (ie, not approved in that country, other than soticlestat), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Note: Compatibility will be determined on the basis of consultation with the sponsor/designee.
2. The participant has a known hypersensitivity to any component of the soticlestat formulation.
3. Participants aged ≥6 years who have positive answers on item numbers 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) before dosing are excluded. This scale will only be administered to participants aged ≥6 years at the time of enrollment or participants who turn 6 after enrollment.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Epilepsihospitalet Filadelfia, Dianalund, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …).

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/289390a307ed459b??page=1&idFilter=TAK-935-3004

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the Sponsor due to a business decision (no safety concerns) as sufficient results were obtained from the previous studies and supplementary data from this study was not required. As there was only 1 participant in this study, no data is reported in order to protect and maintain participant privacy/confidentiality.
Groups:
- Soticlestat: Participant received soticlestat at a starting dose of 100 milligrams (mg) to 200 mg in the 4-week titration. As a part of maintenance (initially planned for 48 weeks per protocol), participant remained on the 200 mg twice daily (BID) dose for 9 days followed by a 1-week taper to receive soticlestat 100 mg BID.
Period: Overall Study
Arm/Group | Soticlestat
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor due to a business decision (no safety concerns) as sufficient results were obtained from the previous studies and supplementary data from this study was not required. As there was only 1 participant in this study, no data is reported in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Soticlestat
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]
Ethnicity (NIH/OMB) [unit: participants]
Race (NIH/OMB) [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Convulsive Seizure Frequency Per 28 Days During First 12 Weeks of Maintenance Period for DS Participants
Time Frame: Baseline to Week 12 of Maintenance Period
Population: as for baseline characteristics
Arm/Group | Soticlestat
Number analyzed (Participants) | 0

2. Primary Outcome: Percent Change From Baseline in Major Motor Drop (MMD) Seizure Frequency Per 28 Days During First 12 Weeks of Maintenance Period for LGS Participants
Time Frame: Baseline to Week 12 of Maintenance Period
Population: as for baseline characteristics
Arm/Group | Soticlestat
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Day 82
Description: The study was terminated by the Sponsor due to a business decision (no safety concerns) as sufficient results were obtained from the previous studies and supplementary data from this study was not required. As there was only 1 participant in this study, no data is reported in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Soticlestat
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT06422377/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT06422377/SAP_001.pdf